CLINICAL TRIAL: NCT01343368
Title: A Phase II Trial of GnRH Agonist for the Preservation of Ovarian Function After Hematopoietic Cell Transplantation (HCT)
Brief Title: Preservation of Ovarian Function After Hematopoietic Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Minnesota Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010LS053; 012M93555 (Other: Institutional Review Board, University of Minnesota)
Record Dates: First submitted 2011-03-15; First posted 2011-04-28 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Multiple Myeloma; Non-Hodgkin Lymphoma; Hodgkin Disease; Acute Myeloid Leukemia; Myeloproliferative Disorders
Keywords: Post-menarchal
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Myeloid, Acute; Myeloproliferative Disorders | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional - Received Leuprolide (Experimental): Long-acting leuprolide 11.25 mg intramuscularly (IM) pre-HCT and 3 months post-HCT PLUS Short-acting leuprolide 0.2 mg subcutaneously (SQ) daily for 14 days for patients who undergo myeloablative allogeneic or autologous hematopoietic cell transplantation.
  Interventions: Drug: Leuprolide; Biological: hematopoietic cell transplant
- Observational Arm (Active Comparator): Women undergoing reduced intensity allogeneic HCT will be observed. Progestin contraceptives, Norethindrone acetate, and any other hormone methods can be used according to the prescription guidelines except for GnRH agonists to suppress menses.
  Interventions: Biological: reduced intensity allogeneic HCT

INTERVENTIONS:
Drug: Leuprolide — Long-acting leuprolide 11.25 mg intramuscularly (IM) pre-transplant (HCT) and 3 months post-HCT PLUS Short-acting leuprolide 0.2 mg subcutaneously (SQ) daily for 14 days
  Other Names: Lupron Depot-3(R); Leuprolide acetate
  Arms: Interventional - Received Leuprolide
Biological: hematopoietic cell transplant — Conventional bone marrow transplant regimen.
  Other Names: HCT
  Arms: Interventional - Received Leuprolide
Biological: reduced intensity allogeneic HCT — A reduced-intensity conditioning transplant is a bone marrow or cord blood transplant (also called a BMT) that uses less intense treatment to prepare for transplant than a standard transplant does. While a standard transplant uses the pre-transplant treatment to destroy most of the disease cells, a reduced-intensity transplant relies on the donor's immune cells to fight disease.
  Other Names: RIC
  Arms: Observational Arm

SUMMARY:
Women undergoing myeloablative allogeneic hematopoietic cell transplant (MA HCT) will receive GnRH agonist leuprolide. Women undergoing reduced intensity allogeneic (RIC) HCT will be observed.

DETAILED DESCRIPTION:
This study is to use gonadotropin releasing hormone (GnRH) agonist leuprolide prior myeloablative hematopoietic cell transplantation to prevent ovarian dysfunction in post-menarchal women.

The primary objective is to determine the effect of GnRH agonists on the incidence of ovarian failure.

The secondary objectives are

* to determine how effective GnRH agonists are at suppressing menses during
* to determine the incidence and timing of resumption of menstrual cycles after HCT
* to determine the incidence and timing of resumption of normal FSH and LH levels after HCT
* to determine the incidence of normal AMH levels after HCT
* to determine the effect of GnRH agonists on immune reconstitution after HCT
* to assess the safety and tolerability of GnRH agonists in the context of HCT

A total of 47 patients will be accrued in this study.

ELIGIBILITY:
Inclusion Criteria:

* Interventional Arm:

  * Eligible for myeloablative allogenic or autologous hematopoietic cell transplant (HCT)
  * Post-menarchal female < or = 50 years of age
  * Normal antimullerian hormone (AMH) level and/or follicle stimulating hormone (FSH)/leuprolide (LH) levels for age/stage of puberty
  * Those women who have an FSH > 40 IU/L and whose diagnosis of malignancy and whose chemotherapy treatment was within 12 weeks of enrollment are still eligible if they had normal menstrual cycles pre-diagnosis.
* Observational Arm:

  * Eligible for reduced intensity allogeneic HCT
  * Post-menarchal female ≤ 50 years of age
  * Normal AMH level and/or FSH/LH for age/stage of puberty
  * Those women who an FSH >40 IU/L and whose diagnosis of malignancy and chemotherapy treatment was within 12 weeks of enrollment are still eligible if they had normal menstrual cycles pre-diagnosis.

Exclusion Criteria:

* All Arms:

  * History of ovarian cancer
  * Surgical resection of one or both ovaries. Prior hysterectomy is allowed as long as the ovaries are intact.
  * Use of GnRH agonist in last 12 months will exclude patients if lab results are not available to demonstrate adequate ovarian function prior to initiation of GnRH therapy.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Smith, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Started | 9 | 10
Completed | 7 | 10
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional - Received Leuprolide | Observational Arm | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 6 | 8
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Number of Patients With Ovarian Failure
Description: Comparison of treatment arms; interventional versus observational. Ovarian failure rate is based on FSH measured at 180 days after HCT; to determine the effect of GnRH agonists on the incidence of ovarian failure (i.e. FSH >40 IU/L) after transplant.
Time Frame: Through Day 180 Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 7 | 10
Participants | 3 | 1

2. Secondary Outcome: Comparison of Number of Patients Who Stopped Menstrual Bleeding
Description: Comparison of treatment arms; interventional versus observational. Count of patients who stopped menstrual bleeding; to determine how the effect of GnRH agonists are at suppressing menses during hematopoietic cell transplant
Time Frame: From Baseline Through Day 365
Population: Five patients on the Interventional arm and 10 patients on the Observational arm were lost to follow-up by Day 365.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 2 | 0
Participants | 2 | 0

3. Secondary Outcome: Comparison of Follicle Stimulating Hormone (FSH) Levels
Description: Comparison of treatment arms; interventional versus observational average FSH levels.
Time Frame: Baseline
Population: Four patients on the Observational arm never had any follow-up FSH levels drawn and were removed from this analysis.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 7 | 6
IU/L | 9.3 (8.0) | 4.4 (1.7)

4. Secondary Outcome: Comparison of Follicle Stimulating Hormone (FSH) Levels
Description: Comparison of treatment arms; interventional versus observational average FSH levels.
Time Frame: Day 100
Population: Four patients on the Observational arm never had any follow-up FSH levels drawn and were removed from this analysis. One patient on the Interventional arm and 7 on the Observational arm were lost to follow-up.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 6 | 3
IU/L | 18.4 (19.5) | 9.1 (12.7)

5. Secondary Outcome: Comparison of Follicle Stimulating Hormone (FSH) Levels
Description: Comparison of treatment arms; interventional versus observational average FSH levels.
Time Frame: Day 180
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 6 | 3
IU/L | 47.0 (40.1) | 4.7 (4.7)

6. Secondary Outcome: Comparison of Follicle Stimulating Hormone (FSH) Levels
Description: Comparison of treatment arms; interventional versus observational average FSH levels.
Time Frame: 1 year
Population: Four patients on the Observational arm never had any follow-up FSH levels drawn and were removed from this analysis. Three patients on the Interventional arm and 8 patients on the Observational arm were lost to follow-up.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 4 | 2
IU/L | 61.5 (97.6) | 48.8 (84.5)

7. Secondary Outcome: Comparison of Follicle Stimulating Hormone (FSH) Levels
Description: Comparison of treatment arms; interventional versus observational average FSH levels.
Time Frame: 2 years
Population: Four patients on the Observational arm never had any follow-up FSH levels drawn and were removed from this analysis. All 7 patients on the Interventional arm and 8 patients on the Observational arm were lost to follow-up.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 0 | 2
IU/L |  | 7.1 (4.6)

8. Secondary Outcome: Comparison of Number of Patients Who Resumed Menstrual Cycles
Description: Comparison of treatment arms; interventional versus observational. Count of patients who resumed menses after hematopoietic cell transplant
Time Frame: Day 365 Post Transplant
Population: Only 6 of the 10 patients that started on the Observational Arm were evaluable. The 2 patients were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 7 | 6
Participants | 2 | 4

9. Secondary Outcome: Comparison of Lutineizing Hormone (LH) Levels
Description: Comparison of treatment arms; interventional versus observational average LH levels during study.
Time Frame: Baseline
Population: Four patients on the Observational arm never had any follow-up LH levels drawn and were removed from this analysis.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 7 | 6
IU/L | 19.8 (30.2) | 6.8 (7.6)

10. Secondary Outcome: Comparison of Luteinizing Hormone (LH) Levels
Description: Comparison of treatment arms; interventional versus observational average LH levels during study.
Time Frame: Day 100
Population: Four patients on the Observational arm never had any follow-up LH levels drawn and were removed from this analysis. One patient on the Interventional arm and 7 on the Observational arm were lost to follow-up.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 6 | 3
IU/L | 2.4 (2.7) | 6.4 (7.7)

11. Secondary Outcome: Comparison of Luteinizing Hormone (LH) Levels
Description: Comparison of treatment arms; interventional versus observational average LH levels during study.
Time Frame: Day 180
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 6 | 3
IU/L | 31.1 (32.0) | 4.3 (3.0)

12. Secondary Outcome: Comparison of Luteinizing Hormone (LH) Levels
Description: Comparison of treatment arms; interventional versus observational average LH levels during study.
Time Frame: 1 year
Population: Four patients on the Observational arm never had any follow-up LH levels drawn and were removed from this analysis. Three patients on the Interventional arm and 8 patients on the Observational arm were lost to follow-up.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 4 | 2
IU/L | 31.9 (36.1) | 27.8 (41.6)

13. Secondary Outcome: Comparison of Leuprolide Hormone (LH) Levels
Description: Comparison of treatment arms; interventional versus observational average LH levels during study.
Time Frame: 2 years
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 0 | 2
IU/L |  | 5.6 (4.3)

14. Secondary Outcome: Comparison of Antimullerian Hormone (AMH) Levels After Transplant
Description: Comparison of treatment arms; interventional versus observational average AMH levels after receiving transplant.
Time Frame: Day Prior to Transplant
Population: Six patients on the Observational arm never had any follow-up AMH levels drawn and were removed from this analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 7 | 4
ng/ml | 0.6 (0.9) | 6.4 (7.7)

15. Secondary Outcome: Comparison of Antimullerian Hormone (AMH) Levels After Transplant
Description: Comparison of treatment arms; interventional versus observational average AMH levels after receiving transplant.
Time Frame: Day 180 after Transplant
Population: Four patients on the Observational and 10 patients on the Observational arm never had any follow-up AMH levels drawn and were removed from this analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Number analyzed (Participants) | 3 | 0
ng/ml | 0.08 (0) |

ADVERSE EVENTS:
Arm/Group | Interventional - Received Leuprolide | Observational Arm
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 3/7 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional - Received Leuprolide (N=7) | Observational Arm (N=10)
Hot Flashes (Vascular disorders) | 3 | 0
Mood Liability (Psychiatric disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No